CLINICAL TRIAL: NCT03395704
Title: A Phase 2, Multi-Center, Randomized, Placebo Controlled, Single-Blind Study With LJPC-401 for the Treatment of Iron Overload in Adult Patients With Hereditary Hemochromatosis
Brief Title: A Study of LJPC-401 for the Treatment of Iron Overload in Adult Patients With Hereditary Hemochromatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LJ401-HH01
Record Dates: First submitted 2017-12-12; First posted 2018-01-10 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Hereditary Hemochromatosis
MeSH Terms: conditions — Hemochromatosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LJPC-401 (Active Comparator): LJPC-401 solution for subcutaneous injection only, 5mg/1 mL (5mg/mL) or 10mg/1mL (10mg/mL) single use vial
  Interventions: Drug: LJPC-401
- Placebo (Placebo Comparator): 0.9% Sodium Chloride Injection, USP, or equivalent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LJPC-401 — LJPC-401 subcutaneous injection, up to 20 mg weekly for 16 weeks. The minimum weekly dose will be 5 mg and the maximum weekly dose of LJPC-401 will be 20 mg.
  Other Names: synthetic human hepcidin
  Arms: LJPC-401
Drug: Placebo — 0.9% Sodium Chloride Injection, USP, or equivalent
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This study is a Phase 2 multicenter, randomized, placebo controlled, single-blind study. The primary objective of the study is to compare the effect of weekly dosing of LJPC-401 (synthetic human hepcidin) versus placebo on transferrin saturation (TSAT) in an adult hereditary hemochromatosis patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical diagnosis of hereditary hemochromatosis
2. Patients who are prescribed therapeutic phlebotomy for treatment of hereditary hemochromatosis
3. Patients with serum ferritin and TSAT levels above treatment guidelines
4. Female patients of child bearing potential must have a negative pregnancy test and must be using a highly effective method of contraception during participation in the study, and for 30 days after the last dose of study drug
5. Males must be surgically sterile (vasectomy), or using a highly effective method of contraception during participation in the study, and for 30 days after the last dose of study drug
6. Patient must be willing and able to provide written informed consent

Exclusion Criteria:

1. Patients receiving iron chelation therapy within 7 days prior to the first dose of study drug
2. Patients initiating phlebotomy treatments less than 3 months prior to the first dose of study drug
3. Pregnant or lactating women
4. Patients taking an immunosuppressive agent without prior Sponsor approval
5. Patients participating in an unapproved investigational drug or investigational therapeutic device within 30 days of study drug
6. Patients who are unwilling or unable to comply with the study protocol requirements
7. Patients with type 1 or poorly controlled type 2 diabetes
8. Patients with a concomitant disease, disability or condition, including laboratory abnormality and ECG findings, which may interfere with the conduct of the study, or which would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this study, including, but not limited to, clinically significant arrhythmias, alcohol dependency or abuse, drug dependency or abuse, or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (18):
  - Investigative Site, North Little Rock, Arkansas
  - Investigative Site, Los Angeles, California
  - Investigative Site, Palo Alto, California
  - Investigative Site, Rialto, California
  - Investigational Site, San Diego, California
  - Investigative Site, San Francisco, California
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Indianapolis, Indiana
  - Investigative Site, Wyoming, Michigan
  - Investigative Site, Jackson, Mississippi
  - Investigative Site, East Setauket, New York
  - Investigative Site, Manhasset, New York
  - Investigative Site, New York, New York
  - Investigative Site, Dallas, Texas
  - Investigative Site, Fort Worth, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Seattle, Washington
- Australia (6):
  - Investigative Site, Liverpool, New South Wales
  - Investigative Site, Westmead, New South Wales
  - Investigative Site, Brisbane, Queensland
  - Investigative Site, Herston, Queensland
  - Investigative Site, Melbourne, Victoria
  - Investigative Site, Murdoch, Western Australia
- France (4):
  - Investigative Site, Bondy
  - Investigative Site, Orléans
  - Investigative Site, Pessac
  - Investigative Site, Rennes
- United Kingdom (3):
  - Investigative Site, Bradford, England
  - Investigative Site, Newcastle upon Tyne, England
  - Investigative Site, Portsmouth, England

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LJPC-401 | Placebo
Started | 34 | 36
Safety Population (The Safety Population included all patients who received at least one dose of study drug.) | 34 | 35
Analysis Population (The Analysis Population included enrolled patients under global protocol Version 4.0 or later, as randomized, who received study drug, and who completed 4 months (Week 16) on study or who had at least 1 phlebotomy after the SOC therapeutic phlebotomy on Day 1 (predose) and before Week 16.) | 21 | 28
Completed | 30 | 33
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | LJPC-401 | Placebo | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 11 | 15 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 18 | 27
  Male | 25 | 17 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 33 | 34 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 35 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 22 | 35
  United Kingdom | 5 | 4 | 9
  Australia | 15 | 7 | 22
  France | 1 | 2 | 3
HH Genotype [Count of Participants; unit: Participants]
  HFE | 1 | 2 | 3
  Not Available | 5 | 5 | 10
  Other | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Effect of LJPC-401 Versus Placebo on Blood Iron Levels
Description: Percentage change in transferrin saturation (TSAT) as measured by blood laboratory tests.
Time Frame: 16 Weeks
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LJPC-401 | Placebo
Number analyzed (Participants) | 21 | 28
Percent Change | -32.8 (20.53) | -2.5 (18.50)
Statistical Analysis 1: Comparison: LJPC-401 vs Placebo; Test type: Superiority; p < 0.0001, General Linear Model

2. Secondary Outcome: Effect of LJPC-401 Versus Placebo on Number of Phlebotomies
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: Phlebotomies
Arm/Group | LJPC-401 | Placebo
Number analyzed (Participants) | 21 | 28
Phlebotomies | 0.52 (0.81) | 2.96 (1.90)

3. Secondary Outcome: Effect of LJPC-401 Versus Placebo on Blood Iron Levels
Description: Change in serum ferritin as measured by blood laboratory tests
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LJPC-401 | Placebo
Number analyzed (Participants) | 21 | 28
Percent Change | -18.0 (25.81) | -18.5 (21.98)

4. Secondary Outcome: Effect of LJPC-401 Versus Placebo on the Total Number of Treatment-emergent Adverse Events
Time Frame: 20 Weeks
Measure: Number; unit: Events
Arm/Group | LJPC-401 | Placebo
Number analyzed (Participants) | 34 | 35
Events | 317 | 101

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | LJPC-401 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/34 | 2/35
Other Adverse Events (participants affected / at risk) | 33/34 | 30/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LJPC-401 (N=34) | Placebo (N=35)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LJPC-401 (N=34) | Placebo (N=35)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (7) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (4) | 5 (5)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 6 (7) | 0 (0)
Injection site erythema (General disorders) | 17 (56) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 2 (7) | 0 (0)
Injection site mass (General disorders) | 3 (7) | 0 (0)
Injection site nodule (General disorders) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 8 (40) | 0 (0)
Injection site pruritus (General disorders) | 14 (50) | 1 (1)
Injection site rash (General disorders) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 4 (29) | 0 (0)
Injection site swelling (General disorders) | 2 (6) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure was restricted for all data, unless published by the company.

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT03395704/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT03395704/SAP_001.pdf